CLINICAL TRIAL: NCT04025541
Title: Analysis of Circulating Tumor Markers in Blood
Acronym: ALCINA2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PROICM 2017-05 BAL
Record Dates: First submitted 2019-06-05; First posted 2019-07-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Breast Cancer; Sarcoma; Lung Cancers; Glioma; Colon Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Sarcoma; Lung Neoplasms; Glioma; Colonic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (13):
- COHORT 1 BREAST TUMOR/PALBOCICLIB (Other): Patient with a locally Advanced tumor or metastatic tumor RH+/HER 2 - , treated by palbociclib
  BLOOD SAMPLING
  Interventions: Biological: Blood sampling
- COHORT 2 BREAST TUMOR / RIBOCICLIB (Other): Patient with a locally Advanced tumor or metastatic tumor RH+/HER 2 - , treated by ribociclib
  BLOOD SAMPLING
  Interventions: Biological: Blood sampling
- COHORT 3 - LUNG CANCER (Other): Patients with histologically proven metastatic bronchial carcinoma eligible for immunotherapy
  Interventions: Biological: Blood sampling C3
- COHORT 4 - CCRm (Other): Patient with metastatic colorectal adenocarcinoma
  Interventions: Biological: Blood sampling C4/7/10/13
- COHORT 5 - T-DXd (Other): Patient with HER2 + metastatic breast cancer, requiring treatment with T-DXd
  Interventions: Biological: Blood sampling C5
- COHORT 6 - Glioma (Other): Patient with grade II, III or IV diffuse glioma
  Interventions: Biological: Blood sampling C6
- COHORT 7 - CIRCUS 2 (Other): Patients with non-metastatic colon cancer
  Interventions: Biological: Blood sampling C4/7/10/13
- COHORT 8 - CTC-AXL Breast (Other): Patients with treatment-naive metastatic breast cancer with distant metastases
  Interventions: Biological: Blood sampling C8
- COHORT 9 - ImmunoTNBC (Other): Patients newly diagnosed with non-metastatic stage II - III early TNBC, requiring neoadjuvant treatment and previously untreated.
  Interventions: Biological: Blood sampling C9
- COHORT 10 - LPS (Other): Patients with well differentiated (WD) liposarcoma, dedifferentiated (DD) liposarcoma or sarcoma other than liposarcoma
  Interventions: Biological: Blood sampling C4/7/10/13
- COHORT 11 - LUNG DRIVER (Other): Patients with Metastatic bronchial carcinoma activating alterations in EGFR (del 19; L858R) or KRAS G12C
  Interventions: Biological: Blood sampling C11 + FFPE
- COHORT 12 - LMD (Other): Patient with breast cancer and suspected with leptomeningeal metastases
  Interventions: Biological: Blood sampling C12
- COHORT 13 - RILA STAB (Other): Patients with breast cancer requiring radiotherapy, whatever the tumor stage
  Interventions: Biological: Blood sampling C4/7/10/13

INTERVENTIONS:
Biological: Blood sampling — blood sampling time : cycle 1 day 15 and cycle 2 day 15 : one sample (6ml) by time
  Other Names: Tumor sampling
  Arms: COHORT 1 BREAST TUMOR/PALBOCICLIB; COHORT 2 BREAST TUMOR / RIBOCICLIB
Biological: Blood sampling C3 — Blood samples will be collected at four key time points:
  * baseline (T1),
  * first scan assessment (T2),
  * second scan assessment (T3),
  * and progression (T4).
  Arms: COHORT 3 - LUNG CANCER
Biological: Blood sampling C4/7/10/13 — Blood samples will be collected before any treatment
  Arms: COHORT 10 - LPS; COHORT 13 - RILA STAB; COHORT 4 - CCRm; COHORT 7 - CIRCUS 2
Biological: Blood sampling C5 — Blood samples will be collected at four key time points:
  * At the inclusion (T1)
  * Before the beginning of the treatment (cycle 1 day 1) (T2)
  * After the first cycle of T-DXd (cycle 2 day 1) (T3)
  * At progression or at the end of the follow-up (after 3 years) (T4)
  Arms: COHORT 5 - T-DXd
Biological: Blood sampling C6 — Blood samples will be collected at three key time points:
  * At the inclusion (T1)
  * For patients starting treatment at the time of inclusion (T2):
  * Chemotherapy: 3 months after inclusion,
  * Concurrent chemoradiotherapy with Temozolomide: 4-6 weeks after completion of radiotherapy,
  * For patients starting treatment at the time of inclusion: at the time of tumor progression if occurring within one year of inclusion, or 12 months after inclusion in the absence of progression (T3).
  Arms: COHORT 6 - Glioma
Biological: Blood sampling C8 — Blood samples will be collected at five key time points:
  * At the inclusion
  * At follow-up visit 2 to 6, every 3 months
  Arms: COHORT 8 - CTC-AXL Breast
Biological: Blood sampling C9 — Blood samples will be collected at four key time points:
  * At the inclusion before the beginning of the treatment (Cycle 1 Day 1)
  * After the first cycle of the first chemo-immunotherapy sequence (Cycle 2 Day 1)
  * After the first cycle of the second chemotherapy sequence (Cycle 2b Day 1)
  * After the end of the whole neo-adjuvant chemo-immunotherapy protocol, before surgery
  Arms: COHORT 9 - ImmunoTNBC
Biological: Blood sampling C11 + FFPE — Blood samples will be collected at five key time points:
  * At the inclusion (T1)
  * At first clinical evaluation (T2): 4th week after start of treatment
  * At first scan evaluation (T3a): 8th week after start of treatment
  * At the Nth scan evaluation (T3b, c, ...)
  * At progression (T4)
  Tumor sampling :
  * At the inclusion
  * At tumor progression
  Arms: COHORT 11 - LUNG DRIVER
Biological: Blood sampling C12 — Blood samples will be collected at several points :
  * Inclusion: at the time of suspected leptomeningeal metastases, prior to any specific treatment,
  * Every 4 weeks until meningeal progression, or for a maximum of 4 months,
  * Then every 3 months beyond 4 months until meningeal progression.
  Arms: COHORT 12 - LMD

SUMMARY:
The circulating tumoral biomarkers in the blood are the object of numerous researches for several decades. The potential clinical interests of these circulating biomarkers are diagnostic, prognostic, predictive of the efficiency of targeted therapies (according to the mutational profile of the cancer), and could allow the study of the mechanisms of resistance under process. In the multiplicity of these blood potential biomarkers joins a permanent evolution of the technological means used to detect them/to quantify, as well as to estimate their clinical utility.

DETAILED DESCRIPTION:
The new major challenge in the research concerns the circulating biomarkers, which aim at replacing the molecular analyses on tumour tissue obtained by biopsy (for example the search for somatic mutations of cancer) by a simple blood test (liquid biopsy). The other current important challenge is to have an idea of the interest to analyse the kinetics of blood markers, in particular in answer to a clinical "event", either through the chemotherapy, a biopsy and / or surgery. There is almost no data in the literature on this aspect. It is very likely that the liberation in the blood of the blood tumoral markers is strongly dependent on medical interventions on the tumour.

The study ALCINA 2 rests exactly on the principle of small cohorts, which correspond each to a clinical situation and/or a technique of different implemented detection, so as to generate data of feasibility and proof of concept. In case of success, statistical hypotheses will be necessary for the implementation of wider studies (being then the object of a specific approval by competent authorities).

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting an invasive tumoral pathology (proved or suspected), whatever is the location or the stage,
2. Man or woman ≥ 18 years,
3. Obtaining of the informed consent signed before any procedure of specific preselection on approval.

Exclusion Criteria:

1. Private persons of freedom or under guardianship,
2. Patient whose regular follow-up is impossible for psychological, family, social or geographical reasons,
3. Pregnant woman and/or breast-feeding,
4. Unaffiliated patient to Social Protection System,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2029-05-29 (Estimated)

PRIMARY OUTCOMES:
Estimation of the feasibility of the various blood tumoral biomarkers analysis | 4 YEARS
  Success rate of the tested detection techniques. The success rate of a given detection technique is calculated by the ratio " detection success " / " number of screened patients"

SECONDARY OUTCOMES:
COHORT 1 and 2 : rate of patients with a grade 3-4 of neutropenia Ciclib-related | 4 YEARS
  Number of participants with treatment-related neutropenia as assessed by CTCAE v4.03
COHORT 1 and 2 : rate of patients with a hepatic toxicity Ciclib-related | 4 YEARS
  Number of participants with treatment-related hepatic toxicity as assessed by CTCAE v4.03
COHORT 3 : Correlation between response to immunotherapy (progressive versus non-progressive) and the number of circulating tumour cells (CTC) expressing the PDL1 marker at T1 (baseline) | 4 years
  Number of CTCs expressing PDL1 at T1
COHORT 4 : To compare the expression of the circulating MS9 mRNA biomarker between healthy subjects and treatment-naive patients with metastatic colorectal cancer | 1 year
  Expression of the MS9 mRNA biomarker
COHORT 5 : to study the impact of baseline HER2+ CTCs detection on PFS under T-DXd treatment | 4 years
  Progression-Free Survival (the primary outcome measure being the HR between CTC+ and CTC- patients, using the HER2+ CTC count at baseline)
COHORT 6 : To develop a computerised procedure for diagnosing glioma based on a nucleoside profile obtained by mass spectroscopy, using Artificial Intelligence | 4 years
  Positive predictive value and negative predictive value of the signature to discriminate glioma vs. no glioma
COHORT 7 : to optimise the culture of circulating tumour cells (CTCs) | 4 years
  Median number of CTCs 1 month after inclusion
COHORT 8 : to evaluate the concordance of CTC-AXL measurement (at inclusion) using the innovative EPIDROP technique and the CellSearch technique | 4 years
  Concordance rate of CTC-AXL measurement (at inclusion) by EPIDROP technique (AXL(-): 0 vs AXL(+): ≥1) and CellSearch technique (AXL(-): 0 vs AXL(+): ≥1)
COHORT 9 : to evaluate the predictive value of circulating immune populations for response to neo-adjuvant chemo-immunotherapy (according to pCR) in patients with early TNBCs, by performing an immunomonitoring before, during and after the treatment. | 4 years
  Response to treatment is defined as a pathological complete response (i.e. no residual invasive tumor in breast and axillary lymph nodes (ypT0ypN0)) after neo-adjuvant therapy.
COHORT 10 : to identify a new non-invasive biological test for the diagnosis of LPS by measuring MDM2 DNA in circulating vesicles | 4 years
  Sensibility and specificity of circulating MDM2 DNA in circulating vesicles for LPS diagnosis
COHORT 11 : to demonstrate a correlation between tumour progression under targeted therapy against EGFR (DEL19; L858R), KRAS G12C and the number of CTCs expressing the HES 1 marker at progression (T4) | 4 years
  Number of CTCs expressing HES 1 to T4
COHORT 12 : to assess the sensitivity of the hepcidin assay in blood for the diagnosis of leptomeningeal metastases of breast cancer, the gold standard being cytological examination of CSF (up to 3 samples). | 4 years
  Sensitivity of the hepcidin value in the 1st blood sample for the diagnosis of leptomeningeal metastases
COHORT 13 : to validate the stability of the RILA at 24hrs (D1), 48hrs (D2), 72hrs (D3) and 96hrs (D4) | 1 year
  The mean RILA at 24h (D1), 48h (D2), 72h (D3) and 96h (D4) will be compared. Equivalences between conditions ((1) 24h and 48h, (2) 24h and 72h, (3) 24h and 96h) will be assessed using Passing & Bablok regression and/or paired t-test. Also, linear regressions between 24h, 48h, 72h and 96h for the same patients will be evaluated in order to determine, if necessary, a conversion formula.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - ICM, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardol T, Eslami-S Z, Masmoudi D, Alexandre M, Duboys de Labarre M, Bobrie A, D'Hondt V, Guiu S, Kurma K, Cayrefourcq L, Jacot W, Alix-Panabieres C. First evidence of AXL expression on circulating tumor cells in metastatic breast cancer patients: A proof-of-concept study. Cancer Med. 2024 Jan;13(1):e6843. doi: 10.1002/cam4.6843. Epub 2023 Dec 22. PMID 38132919
- [Background] Leenhardt F, Fiteni F, Gauthier L, Alexandre M, Guiu S, Firmin N, Pouderoux S, Viala M, Lossaint G, Gautier C, Mollevi C, Gracia M, Gongora C, Mbatchi L, Evrard A, Jacot W. Pharmacokinetic Variability Drives Palbociclib-Induced Neutropenia in Metastatic Breast Cancer Patients: Drug-Drug Interactions Are the Usual Suspects. Pharmaceutics. 2022 Apr 11;14(4):841. doi: 10.3390/pharmaceutics14040841. PMID 35456675
- [Background] Leenhardt F, Alexandre M, Guiu S, Pouderoux S, Beaujouin M, Lossaint G, Philibert L, Evrard A, Jacot W. Impact of pharmacist consultation at clinical trial inclusion: an effective way to reduce drug-drug interactions with oral targeted therapy. Cancer Chemother Pharmacol. 2021 Oct;88(4):723-729. doi: 10.1007/s00280-021-04331-0. Epub 2021 Jul 20. PMID 34286354
- [Background] Leenhardt F, Gracia M, Perrin C, Muracciole-Bich C, Marion B, Roques C, Alexandre M, Firmin N, Pouderoux S, Mbatchi L, Gongora C, Jacot W, Evrard A. Liquid chromatography-tandem mass spectrometric assay for the quantification of CDK4/6 inhibitors in human plasma in a clinical context of drug-drug interaction. J Pharm Biomed Anal. 2020 Sep 5;188:113438. doi: 10.1016/j.jpba.2020.113438. Epub 2020 Jun 22. PMID 32623316